CLINICAL TRIAL: NCT02317393
Title: A Prospective,Multicenter, Phase II Study to Evaluate the Contribution of the Imaging TEP to the Expression of intégrines αvβ3 for the Characterization of the Residual Masses of Non-seminoma Tumors at the End of Chemotherapy
Brief Title: Contribution of the Imaging to the Expression of intégrines αvβ3 for the Characterization of Residual Masses of Non-seminoma Tumors at the End of Chemotherapy
Acronym: TERMATEP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Francois Baclesse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TERMATEP
Record Dates: First submitted 2014-08-25; First posted 2014-12-16 (Estimated); Last update posted 2020-07-09 (Actual); Status verified 2020-02

CONDITIONS: Non-seminomatous Germ Cell Tumors; Metastasis
Keywords: Nuclear medicine; Positron emission tomography; avb3 integrin expression
MeSH Terms: conditions — Nonseminomatous germ cell tumor; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- K5-RGD PET + FDG (Other): Both PET examinations will be performed within 4-6 weeks after the end of chemotherapy, with a maximal delay from end of chemotherapy of 2 months. Delay between FDG and 18F-K5-RGD PET scans will not exceed 2 weeks.
  Interventions: Other: K5-RGD PET; Other: FDG

INTERVENTIONS:
Other: K5-RGD PET — Both PET examinations will be performed within 4-6 weeks after the end of chemotherapy
Other: FDG — Both PET examinations will be performed within 4-6 weeks after the end of chemotherapy

SUMMARY:
The purpose of this study is to evaluate the contribution of the imaging to the expression of intégrines αvβ3 for the characterization of the residual masses of non-seminoma tumors at the end of chemotherapy.

The investigators hope that the results of this first stage of the clinical trial come to consolidate the preclinical results obtained by the investigators team to characterizing the interest and the strong contribution of the use of a tracer resting on the expression of αvβ3 integrine for the diagnosis of simple necrosed mass at the end of the treatment of a non-seminoma tumor, so allowing to defer a surgery to about 40 % of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman aged 18 years or more
* Patients with one or several ganglionic or visceral residual masses (> to 1 cm) after chemotherapy for metastatic non-seminoma testicular tumor, and for which or which a surgery is planned;
* Affiliate to a social security system;
* Signed written Informed consent

Exclusion Criteria:

* Patient deprived of liberty as a result of a justice or administrative decision
* Any medical or psychological condition which could compromise the capacity of the patient to participate in the study;
* Previous or concomitant other cancer in 5 years except basal cell carcinomas

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-12; Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Proportion of teratoma | up to 6 weeks
  Efficacity to differentiate mature teratoma and necroses within the residual masses of germinal non-seminoma tumors.

SECONDARY OUTCOMES:
Metabolic profile | up to 10 weeks
  Number of patients having at least a tumor detected by TEP K5-RGD requiring a surgery, divided by the number of patients having actually at least a tumor (by anatomopathologie) requiring a chirurgie

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas AIDE, Dr, Principal Investigator — Centre François Baclesse, CAEN, France; Arnaud DOERFLER, Dr, Principal Investigator — CHU Côte de Nacre, CAEN, France; Pierre VERA, Dr, Principal Investigator — Centre Henri Becquerel, ROUEN, France
Locations (5):
- France (5):
  - CHU, Caen
  - Centre François Baclesse, Caen
  - Centre Henri Becquerel, Rouen
  - CHU Rouen, Rouen
  - Institut Claudius Regaud, Toulouse